CLINICAL TRIAL: NCT05841030
Title: A Study of Disease Characteristics and Real-life Standard of Care Effectiveness in Patients With Major Depressive Disorder (MDD) With Anhedonia and Inadequate Response to Current Antidepressant Therapy Including an SSRI or SNRI
Brief Title: A Study in Participants With Major Depressive Disorder (MDD) With Anhedonia and Inadequate Response to Current Antidepressant Therapy Including a Selective Serotonin Reuptake Inhibitor (SSRI) or Serotonin Norepinephrine Reuptake Inhibitor (SNRI)
Acronym: VENTURA-RWE
Status: Active, not recruiting | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109332; 67953964MDD3004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MDD Participants With Anhedonia: Data will be collected, for major depressive disorder (MDD) participants with anhedonia who have had an inadequate response to a standard of care (SOC) antidepressant treatment, from participant's source medical records from routine clinical practice over a period of 12 months.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no interventional treatment administered to the participants as a part of this study.

SUMMARY:
The purpose of this study is to assess the socio-demographic, disease-related and treatment-related characteristics, and the standard of care (SOC) treatment patterns of participants with major depressive disorder (MDD) with anhedonia with inadequate response to their current antidepressant treatments and treated according to the standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for single episode or recurrent major depressive disorder (MDD) without psychotic features, according to either the tenth revision of the International Statistical Classification of Diseases and Related Health Problems (ICD-10) or the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Is considered to suffer from a moderate or severe depressive syndrome, as defined by a Montgomery-Asberg Depression Rating Scale (MADRS) total score greater than or equal to (>=) 22 at entry
* Is initiating or is planning to initiate a new add-on antidepressant treatment per local prescribing information to treat the current depressive episode. In the context of this observational study, a new add-on antidepressant treatment is considered any new pharmacological or non-pharmacological treatment that is prescribed in addition to the current antidepressant treatment, inclusive of an selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI or SNRI) with the intent to improve a participant's clinical depressive syndrome. Accordingly, any dose escalation of an antidepressant prescribed prior to baseline or the addition of any drug intended to increase the plasma-concentration of an antidepressant prescribed prior to baseline is not considered a new antidepressant treatment; In parallel with the inclusion of participants considered for add-on strategy, in the United States only, a cohort of approximately 50 participants who switch to a new single (monotherapy) pharmacological antidepressant agent of any antidepressant class per local prescribing information to replace the current antidepressant treatment (that is, "monotherapy switch strategy") will be enrolled. The enrollment of participants with switch to monotherapy will be monitored, and sites will be notified by the sponsor once the planned number for the cohort is achieved. Thereafter, only add-on strategy participants will be enrolled
* Must be capable of providing informed consent (for example, able to read and write), based on the opinion of the participating physician. Must sign (or their legally acceptable representative) an informed consent form indicating that he or she understands the purpose of the study and that he or she agrees to have their data collected and analyzed, in accordance with local requirements and the study protocol
* Meets the criterion for inadequate response to a current antidepressant treatment that includes an SSRI or SNRI (monotherapy SSRI, monotherapy SNRI, combination of antidepressants that includes SSRI/SNRI or SSRI/SNRI augmentation), administered at an adequate dose (as defined in the Massachusetts General Hospital - Antidepressant Treatment Response Questionnaire [MGH ATRQ]) and duration (at least 6 weeks) in the current episode of depression

Exclusion Criteria:

* Has a current or prior diagnosis of a psychotic disorder, MDD with psychotic features, bipolar or related disorders or intellectual disability, according to DSM-5 or ICD-10
* Participants who require an antidepressant (SSRI/SNRI) change (switch to another antidepressant monotherapy), except for a limited number of participants to be recruited in the United States only
* Unstable general medical condition (for example, cardiovascular, respiratory, gastrointestinal, neurologic, hematologic, rheumatologic, immunologic, or endocrine disorders) in the past 3 months that would compromise participation and normal routine medical care per the physician's clinical judgment
* Has lack of treatment response to the current antidepressant therapy that includes a SSRI/SNRI (that is, no [0%] symptomatic improvement despite adequate dose and duration of the antidepressant treatment) assessed using the MGH ATRQ
* History of dementia or mild cognitive impairment. Physician's clinical judgment should document that participant is capable of complying with observational study requirements and being able to complete the appropriate scales
* Has homicidal ideation/intent or is at imminent risk of suicide per the physician's clinical judgment and/or based on the Columbia Suicide Severity Rating Scale (C-SSRS) corresponding to a response of "Yes" on Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consists of participants with MDD with anhedonia who have had an inadequate response to an antidepressant.
Sampling Method: Non-Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Different Socio-demographic Characteristics | Day 1
  Distribution of participants with different demographic characteristics will be assessed.
Percentage of Participants with Disease-related Characteristics | Day 1
  Percentage of participants with disease-related characteristics which includes diagnosis/ disease history and psychiatric/ general medical comorbidities, will be reported.
Percentage of Participants With Type of Therapies and Treatment Strategies | Day 1
  Percentage of participants with type of therapies (such as augmentation, combination therapy, etc.) and treatment strategies will be reported.
Time to Next Antidepressant Treatment | Up to 12 months
  Time to next antidepressant treatment will be reported.
Percentage of Participants with Recurrence or Relapse | Up to 12 months
  Percentage of participants with recurrence or relapse will be reported.
Change From Baseline in Changes in Sexual Functioning Questionnaire (CSFQ-14) Total Score | Baseline, up to 12 months
  Change from baseline in CSFQ-14 total score will be reported. The CSFQ-14 is a structured, self-reported questionnaire designed to measure illness- and medication-related changes in sexual functioning consisting of 14 items that measure sexual functioning as a total score (14 items). Each question rated on a 5-point scale from 1 to 5 with a total score range from 14 to 70. Higher scores reflect higher sexual functioning.
Percentage of Participants With Patient Global Impression of Severity (PGI-S) Scale Score for Sexual Functioning | Up to 12 months
  Percentage of participants with PGI-S scale score for sexual functioning will be reported. The PGI-S is a self-administered, single item questionnaire measuring patients' impression of disease severity. Participants will be asked to rate their disease severity using the following 5-point scale: 1 = None, 2 = Mild, 3 = Moderate, 4 = Severe, and 5 = Very severe. Higher scores indicate greater disease severity.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (95):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham, Homewood, Alabama
  - ATP Clinical Research, California City, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Flagler Hospital and Florida Center for TMS, Saint Augustine, Florida
  - Center for Revitalizing Psychiatry, Sarasota, Florida
  - Interventional Psychiatry of Tampa Bay, Tampa, Florida
  - Atlanta Behavioral Research, LLC, Atlanta, Georgia
  - Psych Atlanta, P.C., Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Baber Research Group, Naperville, Illinois
  - Lumin Health, Newton, Massachusetts
  - Univeristy of Massachusetts, Worcester, Massachusetts
  - Missouri University Health Care South Providence Psychiatry, Columbia, Missouri
  - Signature Research Associates Inc., Fairlawn, Ohio
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Seattle Neuropsychiatric Treatment Center, Tacoma, Washington
- Argentina (7):
  - Fundacion para el Estudio y Tratamiento de las Enfermedades Mentales, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Fleni, Ciudad Autonoma Buenos Aires
  - CEN Consultorios Especializados en Neurociencias, Córdoba
  - Instituto Medico DAMIC, Córdoba
  - Centro Medico Luquez, Córdoba
  - Resolution, Mendoza
- Brazil (5):
  - Hospital Sao Vicente de Paulo, Passo Fundo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, Sao Jose Rio Preto
  - Centro Integrado Facili, São Bernardo do Campo
  - Clinica Viver - Centro de Desospitalizacao Humana, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Canada (5):
  - The Medical Arts Health Research Group, West Vancouver, British Columbia
  - Providence Care Hospital, Kingston, Ontario
  - Introspect Clinic, Ontario, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Jodha Tishon Inc., Toronto, Ontario
- France (9):
  - CHU Angers - Hopital Hotel Dieu, Angers
  - CHU Clermont-Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand
  - Cabinet Medical des Drs Prizac-Desbonnet Scottez, Douai
  - CHU de Grenoble - Hôpital Sud, Isere
  - Hopital la Colombiere, Montpellier
  - CHU de Nantes hotel Dieu, Nantes
  - Cabinet De Psychiatrie Neurostim, Paris
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hopital Sainte Musse, Toulon
- Germany (10):
  - Universitaetsklinikum der RWTH Aachen, Aachen
  - Praxis Dr. med. Kirsten Hahn, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Universitatsklinikum Jena, Jena
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
  - Pharmakologisches Studienzentrum Chemnitz GmbH, Mittweida
  - Gemeinschaftspraxis Prof. Steinbach und Dr. Steib, Nuremberg
  - Praxis Kuehn, Oranienburg
  - Praxis Dipl.-med. Stefan Kusserow, Stralsund
- Italy (9):
  - ASL ROMA, Colleferro
  - Ospedale Policlinico San Martino IRCCS, Genova
  - AUSL LE di Lecce, Lecce
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Pad. Marcora, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Universita degli Studi di Perugia, Perugia
  - Policlinico Tor Vergata, Roma
  - University of Siena, Siena
- South Korea (8):
  - Kyungpook National University Hospital, Daegu
  - CHA University ilsan Medical Center, Goyang
  - Gachon University Gil Medical Center, Incheon
  - Jeju National University Hospital, Jeju Special
  - Kangbuk Samsung Hospital, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (10):
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Gral. de Villalba, Collado Villalba
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Univ. Infanta Leonor, Madrid
  - Csm Fuencarral, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. El Bierzo, Ponferrada
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. Prov. de Zamora, Zamora
- Sweden (4):
  - Gustavsbergs Vardcentral, Gustavsberg
  - Affecta Pskyiatrimottagning, Halmstad
  - ProbarE i Lund AB, Lund
  - ONE LIFETIME Lakarmottagning, Skövde
- United Kingdom (10):
  - Abraham Cowley Unit, Chertsey
  - Kingsway Hospital, Derby
  - Wonford House Hospital, Exeter
  - Kings College Hospital, London
  - Greater Manchester Mental Health NHSFT, Manchester
  - Cumbria, Northumberland, Tyne and Wear NHS Foundation Trust, Newcastle upon Tyne
  - Lincolnshire Partnership NHS Foundation Trust (LPFT), Sleaford
  - Moorgreen Hospital, Southampton
  - St Georges Hospital, Stafford
  - South West Yorkshire Trust, Wakefield

IPD SHARING:
Plan to Share IPD: No